CLINICAL TRIAL: NCT00921843
Title: Methadone in Pediatric Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Evan Kharasch, Vice-Chair for Innovation, Director of Research Entrepreneurship, Duke University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-1195
Record Dates: First submitted 2009-06-10; First posted 2009-06-16 (Estimated); Results first posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-04

CONDITIONS: Anesthesia
Keywords: Pediatric patients undergoing surgery
MeSH Terms: interventions — Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Methadone 0.1mg/kg (Experimental): Methadone 0.1mg/kg
  Interventions: Drug: Methadone 0.1mg/kg
- Methadone 0.2mg/kg (Experimental): Methadone 0.2mg/kg
  Interventions: Drug: Methadone 0.2mg/kg
- Methadone 0.3mg/kg (Experimental): Methadone 0.3mg/kg
  Interventions: Drug: Methadone 0.3mg/kg
- Control (Placebo Comparator): No methadone
  Interventions: Drug: Methadone 0.2mg/kg; Drug: Control

INTERVENTIONS:
Drug: Methadone 0.1mg/kg — Subjects will receive methadone as their intraoperative opioid.
  Arms: Methadone 0.1mg/kg
Drug: Methadone 0.2mg/kg — Subjects will receive methadone as their intraoperative opioid.
  Arms: Control; Methadone 0.2mg/kg
Drug: Methadone 0.3mg/kg — Subjects will receive methadone as their intraoperative opioid.
  Arms: Methadone 0.3mg/kg
Drug: Control — Subjects will not receive methadone as their intraoperative opioid.
  Arms: Control

SUMMARY:
This study will determine the pharmacokinetics of intravenous (IV) methadone in children undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-18
* Undergoing General anesthesia and surgery with anticipated postoperative inpatient stay of greater than or equal to 3 days
* Signed, written, informed consent from legal guardians and assent from patient

Exclusion Criteria:

* History of or known liver or kidney disease

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Kharasch, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Subjects do not receive methadone as their intraoperative opioid.
Period: Overall Study
Arm/Group | Methadone 0.1mg/kg | Methadone 0.2mg/kg | Methadone 0.3mg/kg | Control
Started | 10 | 10 | 11 | 30
Completed | 10 | 10 | 11 | 30
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methadone 0.1mg/kg | Methadone 0.2mg/kg | Methadone 0.3mg/kg | Control | Total
Number analyzed (Participants) | 10 | 10 | 11 | 30 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 10 | 11 | 30 | 61
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 9 | 21 | 42
  Male | 2 | 6 | 2 | 9 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 11 | 30 | 61

OUTCOME MEASURES:

1. Primary Outcome: R-methadone Plasma AUC 0-96hr/Dose
Time Frame: 96 hr
Measure: Mean (Standard Deviation); unit: (ng * hr-1 * ml-1 * mg-1
Arm/Group | Methadone 0.1mg/kg | Methadone 0.2mg/kg | Methadone 0.3mg/kg | Control
Number analyzed (Participants) | 10 | 10 | 11 | 30
(ng * hr-1 * ml-1 * mg-1 | 228 (164) | 189 (54) | 205 (102) | 0 (0)
Statistical Analysis 1: Comparison: Methadone 0.1mg/kg vs Methadone 0.2mg/kg vs Methadone 0.3mg/kg; Test type: Superiority; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 4 days
Groups:
- Methadone 0.1mg/kg: Methadone administration 0.1mg/kg
  Methadone: Subjects will receive methadone as their intraoperative opioid.
- Methadone 0.2mg/kg: Methadone administration 0.2mg/kg
  Methadone: Subjects will receive methadone as their intraoperative opioid
- Methadone 0.3g/kg: Methadone administration 0.3 mg/kg
  Methadone: Subjects will receive methadone as their intraoperative opioid
- Control: No methadone
  No methadone: Subjects will not receive methadone as their intraoperative opioid
Arm/Group | Methadone 0.1mg/kg | Methadone 0.2mg/kg | Methadone 0.3g/kg | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/11 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11 | 0/30
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes